CLINICAL TRIAL: NCT06128161
Title: Comparison of Unilateral CI vs. Bimodal Stimulation in Prosodic Perception
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: 307417
Record Dates: First submitted 2023-09-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hearing Aid — Contralateral Hearing Aid to Cochlear Implant

SUMMARY:
An observational study to determine and assess perception of prosodic information in adults who use bimodal stimulation (cochlear implant plus hearing aid) when using both devices vs. cochlear implant alone.

DETAILED DESCRIPTION:
People with severe to profound hearing loss often do not get satisfactory benefit from their hearing aids. A cochlear implant (CI) is a prosthetic device for the inner ear which can directly stimulate the auditory nerve, bypassing damaged inner ear hair cells and thus provide audible sensations to profoundly deaf patients.

Currently, one CI is funded by NHS England for adult patients and the eligibility criteria for implantation has been relaxed in recent years. As a result, there are now an increasing number of unilateral CI users who possess low-frequency residual hearing in their non-implanted ear. For many patients this residual hearing may still be usefully amplified by a HA. This configuration, consisting of a CI and a contralateral HA, is known as bimodal stimulation.

The PEPS-C receptive test battery has been previously used to assess prosody perception in hearing loss.

The current project will use selected tests from the PEPS-C prosodic test battery to assess intonation, emotion and phrase stress perception ability in adults with bimodal stimulation using both devices together and CI alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Has unilateral Cochlear Implant
* Consistent use of Hearing Aid
* Obtains some benefit in speech discrimination from hearing aid (> 20% AB words)
* Post-lingually deafened
* Fluent English

Exclusion Criteria:

* Longstanding significant asymmetry (> 20 dB HL 4 frequency average) in hearing where the unimplanted ear is the worse ear
* Inconsistent Hearing Aid use
* Significant conductive hearing loss (> 20 dB HL 4 frequency average)
* Using Electro-Acoustic stimulation Cochlear Implant
* Aetiology of hearing loss likely associated with auditory neuropathy
* Significantly abnormal appearance of cochlea or cochlear nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at St. Thomas' Hearing Implant Centre
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
PEPS-C speech test battery | Tested at one time point at day 1 of study after recruitment in both Cochlear Implant Alone and Cochlear Implant and Hearing Aid Together conditions
  Test battery of 7 speech tests examining prosodic elements of speech, each section scored out of 16 (112 in total higher scores better outcome)

SECONDARY OUTCOMES:
AB words speech test | Tested at one time point at day 1 of study after recruitment in both Cochlear Implant Alone and Cochlear Implant and Hearing Aid Together conditions
  Word speech discrimination test in quiet, 30 words presented, scored as % correct, higher score better outcome
SSQ12 Questionnaire | Tested at one time point at day 1 of study after recruitment in both Cochlear Implant Alone and Cochlear Implant and Hearing Aid Together conditions
  Speech Spatial Qualities patient reported outcome measure, scored out of 120 higher scores better outcome
Unaided Soundfield Audiometry | Tested at one time point at day 1 of study after recruitment
  Soundfield hearing test without Cochlear Implant or Hearing Aid
BKB sentences speech test | Tested at one time point at day 1 of study after recruitment in both Cochlear Implant Alone and Cochlear Implant and Hearing Aid Together conditions
  Sentences speech discrimination test in quiet, 100 words presented, 50 male, 50 female voice, scored as %

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom